CLINICAL TRIAL: NCT06973343
Title: Sintilimab Plus Bevacizumab and Chemotherapy on Treatment in Patients With Advanced no Liver Metastatic MSS/pMMR Colorectal Cancer: Phase II Cohort Study
Brief Title: Sintilimab Plus Bevacizumab and Chemotherapy in MSS/pMMR Colorectal With no Liver Metastasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Gang Wang, chief physician, Anhui Provincial Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025004
Record Dates: First submitted 2025-02-21; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who have not received systematic treatment in the past (Experimental): Sintilimab 200mg+ Bevacizumab 7.5mg/kg+Oxaliplatin 130mg/m2+Capecitabine 1250mg/m2 for 6-8cycles, Sintilimab 200mg+ Bevacizumab 7.5mg/kg+Capecitabine 1250mg/m2 as maintenance treatment until disease progression or intolerable toxic side effects occur
  Interventions: Drug: Group A
- Patients who have received first-line systemic treatment in the past (Experimental): Sintilimab 200mg+ Bevacizumab 7.5mg/kg+Irinotecan 150mg/m2+Capecitabine 1250mg/m2 for 6-8cycles, Sintilimab 200mg+ Bevacizumab 7.5mg/kg+Capecitabine 1250mg/m2 as maintenance treatment until disease progression or intolerable toxic side effects occur
  Interventions: Drug: Group B

INTERVENTIONS:
Drug: Group A — Sintilimab 200mg Bevacizumab 7.5mg/kg Oxaliplatin 130mg/m2 Capecitabine 1250mg/m2
  Other Names: Untreated
  Arms: Patients who have not received systematic treatment in the past
Drug: Group B — Sintilimab 200mg Bevacizumab 7.5mg/kg Irinotecan 150mg/m2 Capecitabine 1250mg/m2
  Other Names: After systematic treatment
  Arms: Patients who have received first-line systemic treatment in the past

SUMMARY:
This is a non-randomized, open-label, single-center clinical trial to evaluate efficacy and safety of sintilimab plus bevacizumab and chemotherapy on treatment in patients with advanced no liver metastatic MSS/pMMR colorectal cancer

DETAILED DESCRIPTION:
The regimen involves 3-week cycles with bevacizumab (7.5 mg/m2 on days 1) and fixed doses of sintilimab (200 mg on day 1) and chemotherapy. The primary endpoint is progression-free survival (PFS). Secondary endpoints are Objective response rate(ORR), Disease control rate(DCR), Overall survival(OS) and quality of life. Adverse events are monitored and graded according to the Common Terminology Criteria for Adverse Events version 4.0.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent before implementing any experimental procedures
2. Over 18 years old
3. Histologically confirmed as colorectal adenocarcinoma without liver metastasis
4. At least one measurable lesion (RECIST 1.1)
5. Satellite stable (MSS) or low instability (MSI-L) or normal expression of DNA mismatch repair genes (pMMR)
6. ECOG PS score is 0-1
7. Progress after initial treatment or standard first-line treatment
8. Have sufficient organ and bone marrow function
9. Expected to survive for more than 3 months
10. Participants must have normal hematological test results, including：

    * absolute neutrophil count (ANC) greater than 1.5 × 109/L
    * hemoglobin greater than 8 g/dL
    * platelet count greater than 80-100 × 109/L
11. Participants' prothrombin time (PT) must be less than 1.5 times the upper limit of normal values, and activated partial thromboplastin time (APTT) must be less than 1.5% of the upper limit of abnormal values
12. Participants must have normal laboratory test results, including：serum creatinine levels less than or equal to 1.5 times the upper limit of the normal reference range, or creatinine clearance rates greater than 50 ml/min
13. For participants without liver metastasis, their alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels must be less than or equal to 2.5 times the upper limit of the normal reference range, and their serum total bilirubin levels must be less than 1.5 times the upper limit of the normal reference range
14. For female subjects of childbearing age, a urine or serum pregnancy test with negative results should be conducted within 3 days prior to the first administration of the study drug (Day 1 of the first cycle)
15. If there is a risk of conception, all subjects must use contraceptive measures with an annual failure rate of less than 1% throughout the entire treatment period until 120 days after the last administration of the study drug
16. The subjects must agree to provide sufficient tumor tissue samples for PD-L1 expression detection

Exclusion Criteria:

1. Known presence of active central nervous system (CNS) metastases and/or cancerous meningitis
2. Microsatellite instability (MSI-H) or loss of expression of DNA mismatch repair genes (dMMR)
3. Currently participating in interventional clinical research treatment, or having received other research drugs or used research instruments for treatment within 4 weeks before the first administration
4. Previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs, or drugs that stimulate or synergistically inhibit T cell receptors
5. Within 2 years prior to the first administration, there has been an active autoimmune disease requiring systemic treatment
6. Imaging shows tumor invasion/infiltration into large blood vessels, or researchers or radiologists assess a tendency towards bleeding
7. Have undergone major surgical treatment within 4 weeks prior to the initial administration of the investigational drug (excluding surgery for biopsy purposes) or are expected to undergo major surgery during the study period
8. Severe unhealed wounds, ulcers, or fractures
9. Undertook minor surgeries within 48 hours prior to the first receipt of the study drug
10. Currently or recently (within 10 days prior to receiving the first dose of the study drug) using aspirin (>325 mg/day) or other known nonsteroidal anti-inflammatory drugs that can inhibit platelet function for 10 consecutive days
11. Currently or recently (within 10 days prior to receiving the first dose of the study drug), using full dose oral or parenteral anticoagulants or thrombolytic agents for treatment for 10 consecutive days
12. There is a genetic tendency for bleeding or coagulation dysfunction, or a history of thrombosis
13. Known allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation
14. Individuals known to be allergic to the active ingredients of the study drug
15. Prior to commencing treatment, the individual has not fully recovered from any toxicity and/or complications caused by any intervention measures (i.e., ≤ grade 1 or baseline, excluding fatigue or hair loss)
16. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive)
17. Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected is greater than the upper limit of normal value in the laboratory of the research center)
18. Pregnant or lactating women
19. The presence of any serious or uncontrollable systemic disease

21. Other situations that the researchers believe are not suitable for inclusion, or other potential risks that are not suitable for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 1 year
  Progression free survival

SECONDARY OUTCOMES:
ORR | up to 24 weeks
  Objective response rate
DOR | up to 24 weeks
  Duration of response
DCR | up to 24 weeks
  Disease control rate
OS | through study completion, an average of 2 year
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui provincial cancer hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
Protecting patient privacy

REFERENCES:
- [Background] Fukuoka S, Hara H, Takahashi N, Kojima T, Kawazoe A, Asayama M, Yoshii T, Kotani D, Tamura H, Mikamoto Y, Hirano N, Wakabayashi M, Nomura S, Sato A, Kuwata T, Togashi Y, Nishikawa H, Shitara K. Regorafenib Plus Nivolumab in Patients With Advanced Gastric or Colorectal Cancer: An Open-Label, Dose-Escalation, and Dose-Expansion Phase Ib Trial (REGONIVO, EPOC1603). J Clin Oncol. 2020 Jun 20;38(18):2053-2061. doi: 10.1200/JCO.19.03296. Epub 2020 Apr 28. PMID 32343640